CLINICAL TRIAL: NCT06622200
Title: The Effects of Mindfulness-based Intervention on Trait Mindfulness, Cognitive Reappraisal, Behavioral Suppression, and Quality of Life Among Patients Undergoing Hemodialysis.
Brief Title: The Effect of Mindfulness on Emotional Regulations Skills and Quality of Life Among Patients on Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 136-2024
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: End-Stage Kidney Disease
Keywords: hemodialysis; Cognitive reappraisal; Behavioral suppression; mindfulness; quality of life
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (Experimental): The standardized, theory based MBI was introduced to the experimental group (Smith, 2005). This 30-minute protocol involves a series of activities, including paying attention to and being aware of breath, body sensations, thoughts, and sounds without judgment. This protocol is a widely recognized and utilized method due to its simplicity and accessibility, making it an ideal choice for this study (Alhawatmeh et al., 2022; Smith, 2005).
  Participants completed three weekly sessions of MBI for five weeks during their hemodialysis treatments (Alhawatmeh et al., 2022). Participants were provided with audio recordings of the MBI protocol, which they could practice during hemodialysis sessions. These recordings were delivered via email and WhatsApp, depending on their preference. This audio recording was developed based on the Smith's protocol by a certified study researcher who had a higher degree in nursing and extensive experience in practicing MBI.
  Interventions: Behavioral: Mindfulness-based Intervention
- Control Group (No Intervention): The control group did not receive any intervention from the researcher.

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — In the present research, the standardized, theory based MBI was introduced to the experimental group (Smith, 2005). This 30-minute protocol involves a series of activities, including paying attention to and being aware of breath, body sensations, thoughts, and sounds without judgment. This protocol is a widely recognized and utilized method due to its simplicity and accessibility, making it an ideal choice for this study.
  Participants in the experimental group completed three weekly sessions of MBI for five weeks during their hemodialysis treatments (Alhawatmeh et al., 2022). Participants were provided with audio recordings of the MBI protocol, which they could practice during hemodialysis sessions. These recordings were delivered via email and WhatsApp, depending on their preference. This audio recording was developed based on the Smith's protocol by a certified study researcher who had a higher degree in nursing and extensive experience in practicing and delivering MBIs.
  Arms: Mindfulness-based intervention

SUMMARY:
The study aims to investigate how mindfulness-based intervention (MBI) impacts trait mindfulness, cognitive reappraisal, expressive suppression and quality of life in patients with end-stage renal disease (ESRD) undergoing hemodialysis.

A Randomized controlled trial will be conducted with patients diagnosed with ESRD and undergoing hemodialysis treatment. Participants selected using a convenience sampling method will be randomly assigned into the intervention group (n=52) who received MBI, and the control group (n=52) who received a similar intervention after the study. The intervention involves a 30-minute MBI introduced three sessions per week during hemodialysis sessions over five weeks. Outcome measures included the Mindful Attention Awareness Scale (MAAS) to assess trait mindfulness, the Emotion Regulation Questionnaire (ERQ) for cognitive reappraisal and behavioral suppression, and the Kidney Disease-related Quality of Life Questionnaire for quality of life. Data were collected at baseline and post-intervention.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a comprehensive term encompassing various stages of diminishing kidney function. Kidney damage or sustained estimated glomerular filtration rate (eGFR) of less than 60 ml/min per 1.73 square meters sustained for three months or more are hallmarks of chronic kidney disease (CKD). Individuals affected by CKD commonly encounter symptoms such as fatigue, headaches, weakness, nausea, vomiting swelling in the legs and feet occurs frequently. Challenges in concentration also manifest. If left untreated, CKD can lead to serious complications such as fluid retention high blood pressure, anemia bone disease. Effective management of CKD, such as regular monitoring, lifestyle changes, medication, and other medical interventions remains pivotal in mitigating its progression and associated complications. Left unaddressed, CKD has the potential to advance to end-stage renal disease (ESRD). This necessitates life-saving interventions like dialysis or kidney transplantation (Khusainova et al., 2023; Vaidya & Aeddula, 2023).

ESRD has emerged as a leading global cause of death, standing out as one of the few non-communicable diseases with a rising mortality rate over the past two decades. Over 800 million people worldwide suffer from ESRD, a degenerative illness that affects more than 10% of the population (Kovesdy, 2022). In the United States, ESRD exhibits an incidence rate of 390.2 cases per million and a prevalence rate of 242 cases per million. Black and Hispanic patients had rates of ESRD that were 3.4 and 1.5 times higher, respectively, then those of the general population. Individuals aged 65 and older are at the highest risk of developing ESRD, accounting for about three-quarters of all cases (Johansen et al., 2021).

The prevalence of chronic kidney disease (CKD) is highest in low- and middle-income nations, where controlling its effects is difficult (Kovesdy, 2022). In Jordan, the Jordanian Ministry of Health (MOH) (2020) states that the total number of patients who were registered and treated in the Jordanian Renal Registry will be 7747 by the end of 2020, of which 7290 are Jordanians (94. 1%) and 457 are non-Jordanians (5.9%). The number of Jordanian patients enrolled and hospitalized for ESRD in 2020 was 7290, while the number of new ESRD cases in 2020 was 975, with 898 (92.1%) Jordanians and 77 (7. 9%) non-Jordanians (Jordanian Ministry of Health, 2020).

Renal replacement therapies become necessary when kidneys can no longer perform essential functions ensuring that waste products and excess fluid are removed from the body adequately (Vaidya & Aeddula, 2023). Among renal replacement therapies, hemodialysis is a key therapy that extends life by excreting or removing harmful waste products of metabolism from the circulatory system of humans. Of patients with ESRD, hemodialysis accounts for 70.7% of treatment, with kidney transplantation accounting for 29.3% of cases in the United States (Johansen et al., 2021). In Jordan, the total number of dialysis machines (944) in all units was distributed as follows: 441 (47%) machines in Ministry of Health units, 86 (9%) machines in Royal Medical Service (RMS) units, 32 (3%) machines in university hospitals, and 385 (41%) machines in private sector hospitals. Of the 7290 patients with prevalent ESRD, 3318 patients (45.5%) were treated in dialysis units of the Ministry of Health, 1424 patients (19.5%) in RMS dialysis units, 191 patients (2.6%) in dialysis unit of the University Hospital, and 2,357 patients (32.3%) were treated in private dialysis units.

Despite its role in extending the lives of patients with ESRD, research indicates that individuals undergoing hemodialysis experience a lower quality of life (QOL) compared to those with other chronic illnesses (Dehghan et al., 2020). QOL is a widely recognized concept that reflects an individual's perception of their physical health, psychological well-being, independence, social relationships, beliefs, and personal values (Madadkar & Basiri, 2018). Patients with ESRD undergoing hemodialysis face numerous physical symptoms that limit their daily functioning and threaten their overall physical health. Also, the treatment itself is physically and mentally demanding, as patients typically receive hemodialysis 2 to 3 times per week for 4 to 5 hours per session, which significantly impacts their psychosocial well-being. The combined effects of the illness and the treatment create a substantial burden, jeopardizing the overall QOL for those undergoing hemodialysis (Lim & Lee, 2022).

Patients on hemodialysis who experience a decline in QOL may experience effects on many aspects of their lives, including a diminished capacity to do daily tasks (Madadkar & Baser, 2018). Furthermore, poor QOL contributes to dependency, sadness, social isolation, a reduction in daily activities, and a rise in the financial burden (Dehghan et al., 2020). The work, familial, and social status of individuals with ESRD also altered because of changes in their quality of life (Adamopoulou et al., 2019; Nguyen et al., 2022) Hence, effectively managing diminished QOL and addressing its underlying symptomatic causes are crucial for enhancing clinical outcomes in individuals undergoing hemodialysis. Both pharmacological and non-pharmacological approaches are employed to address these issues. However, a significant number of patients continue to experience psychosomatic symptoms even with the utilization of medications. Presently, there is a growing focus on integrating non-pharmacological and complementary therapies within healthcare systems for improved outcomes (Madadkar & Basiri, 2018). Methods in complementary medicine typically carry minimal side effects and risks, making them suitable for standalone use or in conjunction with other approaches (Kaplan Serin et al., 2020). These therapies, known for their holistic nature, are employed to enhance both the physical and mental well-being of patients (Nguyen et al., 2022).

Mindfulness-based intervention (MBI) is a common and effective complementary therapy that has widespread use in a variety of contexts, groups, and applications (Howarth et al., 2019). MBI teaches people how to cultivate a non-judgmental awareness that is oriented toward the present moment. This intervention has shown potential for treating a number of mental health conditions, including anxiety and depression, as well as persistent physical illnesses (Rigas et al., 2022). In hemodialysis settings, MBI has been found to be effective in improving multiple psychosomatic symptoms such as perceived stress, emotion regulation, sleep disturbances, stress, depression, and anxiety in patients with ESRD worldwide (Razzera et al., 2021). Also, there is initial evidence in the literature supporting the beneficial effect of MBI on quality of life in such patients (Alhawatmeh et al., 2022).

There have been several studies supporting the potential positive effects of MBI on psychophysical health and overall QOL among patients undergoing hemodialysis. However, the mechanisms underlying the beneficial effects of MBI on health among such patients have been rarely studied. In recent years, there has been an increasing interest in identifying the underlying mechanisms of MBI because of growing evidence of its benefits on mental disorders and physical well-being (Gu & Zhu, 2022; Zhang et al., 2021). Several theoretical approaches have been suggested to identify how MBI affects quality of life.

The mechanisms of MBIs have been hypothesized to involve improvements in trait mindfulness, which then facilitate gains in emotion regulation skills, thereby culminating in improved quality of life outcomes (Niazi & Adil, 2017; Shapero et al., 2018; Teper & Inzlicht, 2013; Zhang et al., 2021). T. Indeed, this view is supported by evidence from several studies (Niazi & Adil, 2017; Shapero et al., 2018; Teper & Inzlicht, 2013; Zhang et al., 2021). In the context of the above-outlined framework, the major two strategies for emotion regulation that are mostly studied include cognitive reappraisal and behavioral suppression. Research showed that MBIs enhance cognitive reappraisal, described as reinterpretation of stressful situations in a positive way to lower emotional distress. Evidence on the effectiveness of MBI in behavioral suppression, understood as the suppression of emotional expressions, remains scant and ambiguous. Though findings might be mixed, some studies do indicate a possible positive influence of MBI on cognitive reappraisal, but when it comes to behavior suppression, their effect is negligible or non-significant. This may be related to the fact that the basic mechanism of MBI tends to improve trait mindfulness through present-moment awareness and acceptance rather than suppression of emotions.

Despite these advances, evidence is still developing, and more research needs to be done in order to understand how MBI relate to disparate strategies for regulating emotions. Importantly, such processes have not as yet been investigated empirically in hemodialysis patients-a population experiencing emotional burdens and low quality of life. To the best of our knowledge, no study has yet systematically investigated how MBI would affect emotion regulation processes, namely cognitive reappraisal and expressive suppression, in this patient population. Furthermore, the wider effects of MBI on trait mindfulness and quality of life among hemodialysis patients remain largely unaddressed. The present study therefore tried to fill these gaps in knowledge by assessing the impacts that MBI have on trait mindfulness, cognitive reappraisal, and expressive suppression in hemodialysis patients. It further aimed to explore the impact of MBI on quality of life, thereby offering insight into possible therapeutic benefits that may be gained from the practice of MBI in this highly specific clinical setting.

Methodology

Design An experimental study with a pretest-posttest, randomized, parallel control group design was employed. Participants who were selected using a convenience sampling method were randomly assigned into the intervention group who received MBI, and the control group who received the similar intervention after the study. The intervention involved 30-minute MBI introduced three sessions per week during hemodialysis sessions over a five-week period. The study data were collected at baseline and the end of the intervention.

Setting and Sample This study was conducted at a military hospital Military in the dialysis department, which contains 58 dialysis machines. In this department, there are three sessions per day throughout the week, with three dialysis sessions for each patient per week. The dialyis department receives approximately 174 patients daily, divided into three sessions throughout the day. This dialysis department is considered as the largest dialysis unit in the Middle East, with a monthly capacity of between 2,200 and 2,240 patients (Shqeirat et al., 2021).

Determination of Sample Size G*power 3.1.9.4 was used to calculate the sample size. Given an independent t-test, a medium effect size of 0.5, an alpha of 0.05, and a power of 0.8, the calculated sample size was 102. Taking in consideration an attrition rate of 15 % (Alhawatmeh et al., 2022), the required sample size is 117 participants. To be more conservative, 3 participants were added, resulting in a final required sample size of 120 participants. Of the 170 assessed for eligibility, 120 participants were deemed eligible and agreed to participate. Of these, 104 completed the study and their data were analyzed. The remaining 16 participants chose to withdraw from the study before baseline data collection due to health issues (See Figure 1).

Intervention In the present research, the standardized, theory based MBI was introduced to the experimental group (Smith, 2005). This 30-minute protocol involves a series of activities, including paying attention to and being aware of breath, body sensations, thoughts, and sounds without judgment. This protocol is a widely recognized and utilized method due to its simplicity and accessibility, making it an ideal choice for this study (Alhawatmeh et al., 2022; Smith, 2005).

Smith's (2005) MBI protocol comprises six components:

The MBI protocol developed by Smith (2005) consists of six parts:

1. Practicing mindfulness of the breath by inhaling deeply and slowly, paying attention to the movement of air.
2. Practicing body awareness by paying attention to all of the senses the body has from head to toe and recording any sensations you experience.
3. Being aware of the thought by paying attention to the mind as ideas and thoughts arise and pass, noting them, letting them go, and returning to the mind again and again.
4. Paying attention to sounds without passing judgment on them, observing them, letting them go, and waiting still are examples of mindfulness of sound.
5. Walking mindfully by visualizing yourself on a road devoid of obstacles. Just picture the location of each step without considering where to go.
6. Full meditation: by opening one's eyes and living mindful of the world of the moment, when noting something (sound, thought, sensation, etc.), the individual must let it go and wait for what comes next.

Participants in the experimental group completed three weekly sessions of MBI for five weeks during their hemodialysis treatments (Alhawatmeh et al., 2022). Participants were provided with audio recordings of the MBI protocol, which they could practice during hemodialysis sessions. These recordings were delivered via email and WhatsApp, depending on their preference. This audio recording was developed based on the Smith's protocol by a certified study researcher who had a higher degree in nursing and extensive experience in practicing and delivering MBIs. The audio recording was validated by two psychologists who have good experience of MBIs. The researcher supervised the delivery of the MBI, manage any interruption and protect privacy during the MBI delivery and make sure they could practice successfully. Participants were encouraged to practice the MBI at home during the five-week study period, although it was not mandatory. Participants in both groups were instructed to maintain their usual routines before the study and to avoid seeking psychiatric or alternative treatments for mood improvement. They were also asked to inform the researcher if they decided to pursue such treatments during the study period.

A face-to-face educational session prior to the intervention was performed in order to enhance participants' understanding of the intervention. Accordingly, there was an additional 2-hour education session in which the participants in the experimental group had detailed information from the researcher regarding the purpose and method of intervention. The session included a thorough walkthrough of the entire intervention process; participants were introduced to the basics of the MBI program. The participants were encouraged to ask questions and engage in discussions to ensure a clear understanding of the intervention. The researcher gave an examples to illustrate the potential outcomes and benefits of the intervention. Overall, the pre-intervention training session aimed to establish a solid foundation of knowledge and create a sense of confidence among the experimental group's participants regarding the intervention's effectiveness and implementation (Alhawatmeh et al., 2022).

The control group did not receive any intervention from the researcher. However, upon completion of the study, the control group participants were provided with and given an explanation of the audio recordings of the intervention protocol.

Procedure After getting the IRB approval, the hospital managers were contacted by a study researcher to obtain approval for conducting the study in their institution. When approved, the researcher contacted patients in person to explain the purpose and procedure of the study. Patients agreeing to participate in the study were requested to sign the informed consent form. Then, the participants randomly allocated into the experimental group and control group using a cluster random assignment to avoid contamination. To conduct this assignment strategy, a list of patients who met the study criteria was compiled, including their shifts (A, B, and C). Patients received their hemodialysis sessions three times per week, either on Sunday, Tuesday, and Thursday (STT), or on Monday, Wednesday, and Saturday (MWS). This setup resulted in six clusters (two shifts per week (STT or MWS) × three shifts (A, B,and C) per day). The clusters were defined based on the combination of hemodialysis days and shifts: 1) STT Shift A, 2) STT Shift B, 3) STT Shift C, 4) MWS Shift A, 5) MWS Shift B, and 6) MMWS Shift C. All six clusters, each comprising 20 participants as determined during the sample size calculation, were first listed. Subsequently, these clusters were randomly assigned to either the experimental group or the control group. Randomization was achieved using a random number generation method to ensure an unbiased allocation. This randomization strategy was performed by an independent researcher who did not participate in the recruitment process and remained blinded to the participant list.

After randomization, the study sociodemographic and dependent variables were measured at baseline in the hemodialysis unit before starting the intervention. At the end of the intervention (after five weeks of the actual MBI training), the study dependent variables were measured again. A well-trained research assistant who would not be involved in other study parts collected the data. This research assistant is an experienced nephrology registered nurse. All measurements were privately taken in similar situations (e.g, sitting position) and environments (e.g temperature) in the hemodialysis unit. Nobody was present when they filled out the questionnaire.

Data Analysis The statistical package for social science (SPSS) version 25 was used to analyze data. Descriptive statistics was used to describe the study data as appropriate. Frequency and percentage was used to describe the categorical variables while mean and standard deviation was used to describe the continuous variables. The assumptions for the t-test were tested to confirm the validity of the study results. Normality was examined using histograms, the Shapiro-Wilk test, and by evaluating skewness and kurtosis values. Homogeneity of variance was checked using Levene's test. These checks ensured that the data sufficiently met the necessary assumptions for performing the t-tests. Independent t-tests was used to examine any baseline differences between the study groups on the continuous sociodemographic variables and main study outcomes. Chai square tests were used to examine any baseline differences between the study groups on the categorical sociodemographic variables. A dependent t-test was used to assess changes in the mean scores of the outcomes between the pre-test and post-test within each study group. Finally, independent t-tests were used to examine the significant differences between the study groups at end of the intervention.

Ethical Considerations The Institutional Review Board (IRB) approved the proposed study (Approval Number: 136-2024). Participants who agreed to participate in the study were asked to sign a consent form that described the purpose and scope of the research. They confirmed that they had the freedom to reject participation in the study and that such rejection would not affect the care they received. They were assured that the research data would be stored in a secure location in a locked cabinet accessible only to the researcher, with numbers replacing their names to avoid their personal identification. No patients were excluded from the trial because of their gender, race, or nationality. During the intervention, if any patient felt dizzy or uncomfortable, the intervention was stopped, and the attending physician was informed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD undergoing hemodialysis at least three sessions a week
* Being at least 18 years old
* Having a smartphone
* Being capable of reading and writing in Arabic

Exclusion Criteria:

* Patients under psychotherapy or taking regular psychopharmacological and analgesic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
kidney Disease- related Quality of Life questionnaire | From enrollment to the end of treatment at 6 weeks
  The Arabic version of the kidney disease- related Quality of Life questionnaire (KDQOL-36) was used to evaluate quality of life. It has four subscales: symptoms and problems (12 items); burden of kidney disease (4 items); effects of kidney disease (8 items); and generic core [Physical Component Summary (PCS, 12 items) and mental component summary (MCS, 12 items) (Elamin et al., 2019). Each item's raw, pre-coded numerical values are converted linearly to a scale from 0 to 100, where higher numbers indicate better quality of life (Kalantar-Zadeh & Unruh, 2005). The Arabic version of the scale revealed favorable psychometric attributes in Arabic patients with chronic renal insufficiency and The KDQOL-36 translation showed a Cronbach's alpha of 0.81, demonstrating strong internal reliability (Alhawatmeh et al., 2022; Elamin et al., 2019).

SECONDARY OUTCOMES:
Emotional Regulation Questionnaire | From enrollment to the end of treatment at 6 weeks
  The Arabic version of the Emotion Regulation Questionnaire (ERQ) developed by Keshky (2018) was used to assess cognitive reappraisal and expressive suppression. The scale consists of 10 items, each rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). The scale consists of two subscales measuring two emotion regulation abilities: expressive suppression (4 items) and cognitive reappraisal (6 items). The higher scores indicate greater emotion regulation abilities (Gross & John, 2003). The Arabic version showed valid and reliable results among Arabic Gulf population and patients undergoing hemodialysis with the Cronbach alpha of the study instrument is 0.83 (Alhawatmeh et al., 2022; Keshky, 2018).
Mindful Attention Awareness Scale | From enrollment to the end of treatment at 6 weeks
  The Mindful Attention Awareness Scale (MAAS) is a widely used self-report measure designed to assess an individual's trait mindfulness-their general capacity to be present and attentive to ongoing experiences in daily life. The MAAS typically consists of 15 items. Patients rate how frequently they experience various characteristics of mindfulness in day-to-day activities. Participants rate each item on a Likert-type scale. This scale indicates frequency of experiences from "1: almost always" to "5: almost never" (Brown & Ryan, 2003). Score ranges from 15 to 75. Higher scores reflect a greater tendency to be mindful and present in daily life. Strong convergent validity and internal consistency are demonstrated by Arabic MAAS among Arab hemodialysis patients (Alhawatmeh et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, Doctoral degree, Principal Investigator — Hossam alhawatmeh, associate professor, Jordan university of science and technology
Locations (1):
- Prince Rashid Military Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Because of ethical restrictions

REFERENCES:
- [Background] Adamoli, A. N., Razzera, B. N., Ranheiri, M. F., Colferai, R. N., Russell, T. A., Noto, A. R., & da Silva de Oliveira, M. (2021). Mindfulness-Based Intervention Performed During Hemodialysis: An Experience Report. Trends in Psychology, 29(2), 320-340. https://doi.org/10.1007/s43076-020-00058-8.
- [Background] Adamopoulou F, Alikari V, Zyga S, Tsironi M, Tzavella F, Giannakopoulou N, Theofilou P. The Effect of Fatigue and Pain Self- Efficacy on Health-Related Quality of Life Among Patients with Multiple Sclerosis. Mater Sociomed. 2019 Mar;31(1):40-44. doi: 10.5455/msm.2019.31.40-44. PMID 31213954
- [Background] Alhawatmeh H, Alshammari S, Rababah JA. Effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in hemodialysis patients: A randomized controlled trial. Int J Nurs Sci. 2022 Mar 8;9(2):139-146. doi: 10.1016/j.ijnss.2022.03.004. eCollection 2022 Apr. PMID 35509694
- [Background] Alhawatmeh HN, Rababa M, Alfaqih M, Albataineh R, Hweidi I, Abu Awwad A. The Benefits of Mindfulness Meditation on Trait Mindfulness, Perceived Stress, Cortisol, and C-Reactive Protein in Nursing Students: A Randomized Controlled Trial. Adv Med Educ Pract. 2022 Jan 13;13:47-58. doi: 10.2147/AMEP.S348062. eCollection 2022. PMID 35046747
- [Background] Alhawatmeh H, Najadat IA, Hweidi IM. Mindfulness-based intervention as a symptom management strategy in patients with end-stage renal disease: A controlled clinical trial. Int J Nurs Pract. 2024 Dec;30(6):e13282. doi: 10.1111/ijn.13282. Epub 2024 Jun 16. PMID 38880954
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Dehghan M, Namjoo Z, Bahrami A, Tajedini H, Shamsaddini-Lori Z, Zarei A, Dehghani M, Ranjbar MS, Rafiee Sarbijan Nasab F. The use of complementary and alternative medicines, and quality of life in patients under hemodialysis: A survey in southeast Iran. Complement Ther Med. 2020 Jun;51:102431. doi: 10.1016/j.ctim.2020.102431. Epub 2020 May 21. PMID 32507442
- [Background] Desrosiers A, Vine V, Klemanski DH, Nolen-Hoeksema S. Mindfulness and emotion regulation in depression and anxiety: common and distinct mechanisms of action. Depress Anxiety. 2013 Jul;30(7):654-61. doi: 10.1002/da.22124. Epub 2013 Apr 16. PMID 23592556
- [Background] Elamin S, E Elbasher AH, E Ali SE, Abu-Aisha H. Arabic translation, adaptation, and validation of the kidney disease quality of life short-form 36. Saudi J Kidney Dis Transpl. 2019 Nov-Dec;30(6):1322-1332. doi: 10.4103/1319-2442.275476. PMID 31929279
- [Background] Fatma, H., Menessy, N., Menessy, R., Ramadan, F., & Kamel, N. (2022). The Relationship between Mindfulness, Emotion Regulation and Mental Well-being among Academic Staff Educators at the Faculty of Nursing. Egyptian Journal of Health Care, 6.
- [Background] Garland EL, Geschwind N, Peeters F, Wichers M. Mindfulness training promotes upward spirals of positive affect and cognition: multilevel and autoregressive latent trajectory modeling analyses. Front Psychol. 2015 Feb 2;6:15. doi: 10.3389/fpsyg.2015.00015. eCollection 2015. PMID 25698988
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Gu YQ, Zhu Y. A randomized controlled trial of mindfulness-based cognitive therapy for body dysmorphic disorder: Impact on core symptoms, emotion dysregulation, and executive functioning. J Behav Ther Exp Psychiatry. 2023 Dec;81:101869. doi: 10.1016/j.jbtep.2023.101869. Epub 2023 May 8. PMID 37311379
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Howarth, A., Smith, J. G., Perkins-Porras, L., & Ussher, M. (2019). Effects of Brief Mindfulness-Based Interventions on Health-Related Outcomes: A Systematic Review. Mindfulness, 10(10), 1957-1968. https://doi.org/10.1007/s12671-019-01163-1.
- [Background] Inker LA, Astor BC, Fox CH, Isakova T, Lash JP, Peralta CA, Kurella Tamura M, Feldman HI. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for the evaluation and management of CKD. Am J Kidney Dis. 2014 May;63(5):713-35. doi: 10.1053/j.ajkd.2014.01.416. Epub 2014 Mar 16. PMID 24647050
- [Background] Johansen KL, Chertow GM, Foley RN, Gilbertson DT, Herzog CA, Ishani A, Israni AK, Ku E, Kurella Tamura M, Li S, Li S, Liu J, Obrador GT, O'Hare AM, Peng Y, Powe NR, Roetker NS, St Peter WL, Abbott KC, Chan KE, Schulman IH, Snyder J, Solid C, Weinhandl ED, Winkelmayer WC, Wetmore JB. US Renal Data System 2020 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2021 Apr;77(4 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2021.01.002. No abstract available. PMID 33752804
- [Background] Kabat-Zinn, J. (1990). Full Catastrophe Living: Using the Wisdom of Your Body and Mind to Face Stress, Pain, and Illness. Dell Publishing.
- [Background] Kaplan Serin E, Ovayolu N, Ovayolu O. The Effect of Progressive Relaxation Exercises on Pain, Fatigue, and Quality of Life in Dialysis Patients. Holist Nurs Pract. 2020 Mar/Apr;34(2):121-128. doi: 10.1097/HNP.0000000000000347. PMID 31567304
- [Background] Keng, S. L., Smoski, M. J., & Robins, C. J. (2011). Mindfulness and Emotion Regulation: Insights from Neuroscience and Clinical Practice. Cognitive Therapy and Research, 35(6), 601-610.
- [Background] Keshky, M. E. E. (2018). Factor Structure, Reliability and Validity of the Arabic Version of the Emotion Regulation Questionnaire (ERQ) in a Sample of Saudi Children and Adolescents. International Journal of Psychology and Behavioral Sciences, 8(2), 22-30.
- [Background] Khusainova, M. A., Khaydarov, S. N., Makhmudova, K. D., & Ortikova, S. X. (2023). Features of prevention of chronic kidney diseases and chronic heart failure. Science and Education, 4(5), Article 5.
- [Background] Kovesdy CP. Epidemiology of chronic kidney disease: an update 2022. Kidney Int Suppl (2011). 2022 Apr;12(1):7-11. doi: 10.1016/j.kisu.2021.11.003. Epub 2022 Mar 18. PMID 35529086
- [Background] Kriakous SA, Elliott KA, Lamers C, Owen R. The Effectiveness of Mindfulness-Based Stress Reduction on the Psychological Functioning of Healthcare Professionals: a Systematic Review. Mindfulness (N Y). 2021;12(1):1-28. doi: 10.1007/s12671-020-01500-9. Epub 2020 Sep 24. PMID 32989406
- [Background] Lee M, Jang KS. Mediating Effects of Emotion Regulation between Socio-Cognitive Mindfulness and Achievement Emotions in Nursing Students. Healthcare (Basel). 2021 Sep 21;9(9):1238. doi: 10.3390/healthcare9091238. PMID 34575012
- [Background] Lee M, Park H. Mediating effects of emotion regulation between socio-cognitive mindfulness and empathy in nurses: a cross-sectional study. BMC Nurs. 2022 Nov 9;21(1):306. doi: 10.1186/s12912-022-01081-z. PMID 36352405
- [Background] Lee, S., & Young, J. (2018). Mind the Gap: The History and Philosophy of Health Psychology and Mindfulness. Revista Psicologia e Saúde, 10, 25. https://doi.org/10.20435/pssa.v10i2.693.
- [Background] A Lim K, Hee Lee J. Factors Affecting Quality of Life in Patients Receiving Hemodialysis. Iran J Public Health. 2022 Feb;51(2):355-363. doi: 10.18502/ijph.v51i2.8688. PMID 35866126
- [Background] Madadkar, & Basiri. (2018). Effect of Relaxation Jacobson on quality of Life and self-efficacy in Patients Undergoing Hemodialysis. Complementary Medicine Journal, 7(4), 2090-2099.
- [Background] Mehrabi, F., & Tavakoli, M. (2022). The Effectiveness of Mindfulness-Based Stress Reduction Intervention for Cognitive Emotion Regulation and Cognitive Reactivity in Patients with Epilepsy. International Journal of Cognitive Therapy, 15(4), 465-478. https://doi.org/10.1007/s41811-022-00144-y.
- [Background] Nguyen SA, Oughli HA, Lavretsky H. Complementary and Integrative Medicine for Neurocognitive Disorders and Caregiver Health. Curr Psychiatry Rep. 2022 Sep;24(9):469-480. doi: 10.1007/s11920-022-01355-y. Epub 2022 Aug 13. PMID 35962927
- [Background] Niazi, S., & Adil, A. (2017). Role of Mindfulness and Psychological Wellbeing Between External Locus of Control and Depression: A Moderated Mediation Model. Peshawar Journal of Psychology and Behavioral Sciences (PJPBS), 3(1), Article 1. https://doi.org/10.32879/pjpbs.2017.3.1.1-19.
- [Background] Razzera BN, Adamoli AN, Ranheiri MF, Oliveira MDS, Feoli AMP. Impacts of mindfulness-based interventions in people undergoing hemodialysis: a systematic review. J Bras Nefrol. 2022 Jan-Mar;44(1):84-96. doi: 10.1590/2175-8239-JBN-2021-0116. PMID 34643641
- [Background] Rigas C, Park H, Nassim M, Su CL, Greenway K, Lipman M, McVeigh C, Novak M, Trinh E, Alam A, Suri RS, Mucsi I, Torres-Platas SG, Noble H, Sekhon H, Rej S, Lifshitz M. Long-term Effects of a Brief Mindfulness Intervention Versus a Health Enhancement Program for Treating Depression and Anxiety in Patients Undergoing Hemodialysis: A Randomized Controlled Trial. Can J Kidney Health Dis. 2022 Mar 4;9:20543581221074562. doi: 10.1177/20543581221074562. eCollection 2022. PMID 35273807
- [Background] Shapero BG, Greenberg J, Pedrelli P, de Jong M, Desbordes G. Mindfulness-Based Interventions in Psychiatry. Focus (Am Psychiatr Publ). 2018 Winter;16(1):32-39. doi: 10.1176/appi.focus.20170039. Epub 2018 Jan 24. PMID 29599651
- [Background] Shqeirat MD, Hijazi BM, Almomani BA. Treatment related problems in Jordanian hemodialysis patients. Int J Clin Pharm. 2021 Oct;43(5):1352-1359. doi: 10.1007/s11096-021-01259-6. Epub 2021 Mar 21. PMID 33748911
- [Background] Smith, J. (2005). Relaxation, meditation, and mindfulness: A mental health practitioner's guide to new and traditional approaches.
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524.
- [Background] Sullivan MJ, Thorn B, Haythornthwaite JA, Keefe F, Martin M, Bradley LA, Lefebvre JC. Theoretical perspectives on the relation between catastrophizing and pain. Clin J Pain. 2001 Mar;17(1):52-64. doi: 10.1097/00002508-200103000-00008. PMID 11289089
- [Background] Teper R, Inzlicht M. Meditation, mindfulness and executive control: the importance of emotional acceptance and brain-based performance monitoring. Soc Cogn Affect Neurosci. 2013 Jan;8(1):85-92. doi: 10.1093/scan/nss045. Epub 2012 Apr 15. PMID 22507824
- [Background] Terkawi AS, Sullivan M, Abolkhair A, Al-Zhahrani T, Terkawi RS, Alasfar EM, Khait SSA, Elkabbani A, Kabbani N, Altirkawi KA, Tsang S. Development and validation of Arabic version of the pain catastrophizing scale. Saudi J Anaesth. 2017 May;11(Suppl 1):S63-S70. doi: 10.4103/sja.SJA_130_17. PMID 28616005
- [Background] Vaidya SR, Aeddula NR. Chronic Kidney Disease. 2024 Jul 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK535404/ PMID 30571025
- [Background] Vaishnav BS, Hirapara JJ, Shah MK. Study of effect of guided meditation on quality of life in patients of end stage renal disease (ESRD) on maintenance hemodialysis - a randomised controlled trial. BMC Complement Med Ther. 2022 Sep 9;22(1):238. doi: 10.1186/s12906-022-03717-8. PMID 36085065
- [Background] Wang YX, Yin B. A new understanding of the cognitive reappraisal technique: an extension based on the schema theory. Front Behav Neurosci. 2023 Apr 17;17:1174585. doi: 10.3389/fnbeh.2023.1174585. eCollection 2023. PMID 37138662
- [Background] Whitfield T, Barnhofer T, Acabchuk R, Cohen A, Lee M, Schlosser M, Arenaza-Urquijo EM, Bottcher A, Britton W, Coll-Padros N, Collette F, Chetelat G, Dautricourt S, Demnitz-King H, Dumais T, Klimecki O, Meiberth D, Moulinet I, Muller T, Parsons E, Sager L, Sannemann L, Scharf J, Schild AK, Touron E, Wirth M, Walker Z, Moitra E, Lutz A, Lazar SW, Vago D, Marchant NL. The Effect of Mindfulness-based Programs on Cognitive Function in Adults: A Systematic Review and Meta-analysis. Neuropsychol Rev. 2022 Sep;32(3):677-702. doi: 10.1007/s11065-021-09519-y. Epub 2021 Aug 4. PMID 34350544
- [Background] WHO | WHOQOL: Measuring Quality of Life. (2020, May 15). https://web.archive.org/web/20200515055014/https://www.who.int/healthinfo/survey/whoqol-qualityoflife/en/.
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] Zhou S, Wu Y, Xu X. Linking Cognitive Reappraisal and Expressive Suppression to Mindfulness: A Three-Level Meta-Analysis. Int J Environ Res Public Health. 2023 Jan 10;20(2):1241. doi: 10.3390/ijerph20021241. PMID 36673984